CLINICAL TRIAL: NCT03882099
Title: Vitamin D Level in Patients With Pre-eclampsia, Eclampsia and Normal Full Term Pregnant
Brief Title: Vitamin D Level and Its Relation to Pre-eclampsia and Eclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yahia El-Faissal, Dr, Cairo University
Other Study IDs: 173019OBGYN
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Vitamin D Deficiency; Pre-Eclampsia; Eclampsia, Antepartum
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant women with pre-eclampsia
  Interventions: Diagnostic Test: Determination of Vitamin D by ELISA
- Pregnant women with eclampsia
  Interventions: Diagnostic Test: Determination of Vitamin D by ELISA
- Normotensive pregnant women
  Interventions: Diagnostic Test: Determination of Vitamin D by ELISA

INTERVENTIONS:
Diagnostic Test: Determination of Vitamin D by ELISA — Blood samples

SUMMARY:
To compare 25(OH)D level in patients with pre-eclampsia, eclampsia and normotensive pregnant women as well as to study the prevalence of Vitamin D deficiency among the 3 groups.

DETAILED DESCRIPTION:
200 patients with pre-eclampsia, 100 with eclampsia and 200 normotensive pregnant controls attending Delivery/emergency department in Kasr Al Ainy hospital will be included in the study (from March 2019 till September 2019). 25(OH) D level will be measured for the three groups.

* Preeclampsia is defined as systolic BP >140 and/or diastolic BP>90 on two occasions, 4 hours apart in pregnant females>20 weeks, plus proteinuria >/= 1+ urine dipstick protein.
* Eclampsia defined as tonic-clonic seizures in women with pre-eclampsia.
* Controls are normotensive pregnant females with no proteinuria and no other medical disorders.
* The determination of 25(OH) D is based on a competitive enzyme-linked immunosorbant assay (ELISA) using the 25(OH)D3/D2 ELISA system (ORGENTIC DIAGNOSTIKA GmbH, Germany)

Inclusion criteria:

Age 20-35 years Gestational age 30-40 weeks

Exclsion criteria:

Twin pregnancy Other medical conditions during prrgnancy Drugs that influence Vit D levels eg.antiepileptics and antituberculous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years
* Gestational age 30-40 weeks

Exclusion Criteria:

* Twin pregnancy
* Other medical conditions during pregnancy
* Drugs that influence Vit D levels eg.antiepileptics and antituberculous treatment

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: 200 patients with pre-eclampsia, 100 with eclampsia and 200 normotensive pregnant controls attending Delivery/emergency department in Kasr Al Ainy hospital will be included in the study
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-17 (Actual); Primary Completion 2019-09-17 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
To compare vitamin D levels in the three groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Publication in journals and presentation in conferences